CLINICAL TRIAL: NCT04108507
Title: Prevention of Residual Low Back Pain After Percutaneous Kyphosis(PKP) Using Posterior Branch Block of Spinal Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, WU YAOSEN, Deputy Director of Spinal surgery, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2018-08-109
Record Dates: First submitted 2019-09-21; First posted 2019-09-30 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Osteoporotic Fracture
Keywords: Percutaneous kyphoplasty（PKP）; nerve block; posterior branch of spinal nerve
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posterior branch block of spinal nerve (Experimental): posterior branch block of spinal nerve during Percutaneous kyphoplasty(PKP)operation
  Interventions: Procedure: posterior branch block of spinal nerve
- without posterior branch block of spinal nerve (No Intervention): without posterior branch block of spinal nerve during Percutaneous kyphoplasty(PKP) operation

INTERVENTIONS:
Procedure: posterior branch block of spinal nerve — posterior branch block of spinal nerve during Percutaneous kyphoplasty(PKP) operation
  Arms: posterior branch block of spinal nerve

SUMMARY:
The purpose of this study was to block the posterior branch of lumbar spinal nerve during PKP operation and compare it with the patients without spinal nerve block, so as to verify the effect of posterior branch block of spinal nerve in relieving short-term and long-term residual low back pain after operation.

DETAILED DESCRIPTION:
Patients older than 60 years old who underwent Percutaneous kyphosis(PKP) surgery for osteoporotic fractures were randomly divided into two groups. The lumbar spinal nerve branch was blocked with betamethasone and ropivacaine in the experimental group during PKP operation, while the lumbar spinal nerve branch block was not performed in the control group during PKP operation. The low back pain was evaluated at 1 week, 2 weeks, 1 month, 3 months and 6 months after operation using Visual analogue pain score(VAS)scale.So as to compare the effect of lumbar spinal nerve block on residual pain after PKP.

ELIGIBILITY:
Inclusion Criteria:

* osteoporotic fracture
* acute vertebral compression fracture (within 2 weeks)
* fracture level lower thanT6

Exclusion Criteria:

* other types of fractures
* patients younger than 60 years of age,
* with other disease (metabolic bone disease, metastasis, uncor- rectable coagulopathy, spinal infection, severe cardiopulmonary comorbidity, cognitive disorders etc)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Residual low back pain after operation | 6 months after operation
  Residual low back pain after operation using Visual analogue pain score(VAS) scale, VAS scores range from 0 to 10, more higher score means more severe pain, and residual back pain was defined as a VAS score greater than or equal to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klazen CA, Lohle PN, de Vries J, Jansen FH, Tielbeek AV, Blonk MC, Venmans A, van Rooij WJ, Schoemaker MC, Juttmann JR, Lo TH, Verhaar HJ, van der Graaf Y, van Everdingen KJ, Muller AF, Elgersma OE, Halkema DR, Fransen H, Janssens X, Buskens E, Mali WP. Vertebroplasty versus conservative treatment in acute osteoporotic vertebral compression fractures (Vertos II): an open-label randomised trial. Lancet. 2010 Sep 25;376(9746):1085-92. doi: 10.1016/S0140-6736(10)60954-3. Epub 2010 Aug 9. PMID 20701962